CLINICAL TRIAL: NCT04508582
Title: Linking the Maternal Immune System to Cardiac Function in Preeclampsia
Brief Title: Cardiac and Immune Cell Function in Preeclampsia
Status: Completed | Type: Observational
Sponsor: Queen Mary University of London (Other)
Collaborators: British Heart Foundation (Other); Barts & The London NHS Trust (Other)
Responsible Party: Sponsor
Other Study IDs: IRAS 281197
Record Dates: First submitted 2020-08-07; First posted 2020-08-11 (Actual); Last update posted 2025-03-10 (Actual); Status verified 2025-03

CONDITIONS: Preeclampsia; Hypertension; Pregnancy Induced Hypertension; Pregnancy Related; Cardiovascular Diseases; Cardiovascular Risk Factor; Heart Diseases
Keywords: Immunology, neutrophil, t-cell, placenta
MeSH Terms: conditions — Pre-Eclampsia; Hypertension; Hypertension, Pregnancy-Induced; Cardiovascular Diseases; Heart Diseases | interventions — Echocardiography; Caves; Hematologic Tests

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Women with Pre-eclampsia: De novo hypertension after 20 weeks gestation with evidence of end organ dysfunction.
  Interventions: Diagnostic Test: Cardiovascular magnetic resonance; Diagnostic Test: Echocardiography; Diagnostic Test: Blood test
- Women with Pregnancy-induced hypertension: De novo hypertension after 20 weeks gestation without evidence of end organ dysfunction.
  Interventions: Diagnostic Test: Cardiovascular magnetic resonance; Diagnostic Test: Echocardiography; Diagnostic Test: Blood test
- Healthy pregnant controls: Low risk women at booking as per NICE guidelines without any medical condition throughout pregnancy
  Interventions: Diagnostic Test: Cardiovascular magnetic resonance; Diagnostic Test: Echocardiography; Diagnostic Test: Blood test

INTERVENTIONS:
Diagnostic Test: Cardiovascular magnetic resonance — Imaging of the heart with CMR, without use of contrast agents.
  Other Names: CMR
Diagnostic Test: Echocardiography — Imaging of the heart with ultrasound.
  Other Names: echo
Diagnostic Test: Blood test — Time- matched blood samples will be taken from patients to assess immune cell phenotype and function, paying particular attention to neutrophil and T-cell phenotype. Plasma samples will be collected for the analyses of cardiac specific factors (BNP, troponin) as well as measurement of steroid hormones (progesterone and oestradiol), and soluble inflammatory and anti-inflammatory mediators

SUMMARY:
Preeclampsia is a multi-system vascular disease which affects 2-5% of pregnancies. It is also a risk factor for the development of cardiovascular disease later in life and a number of functional and structural cardiac changes have been found in this population of patients.

In mouse models disruption of a group of immune cells, neutrophils, has led to alteration of the placenta and offspring consistent with those seen in preeclampsia. These mice also have an abnormal cardiac function and structure (Nadkarni et al 2016). The investigators hypothesis that this may also occur in humans.

This study aims to intimately link the maternal immunological and vascular components of cardiac dysfunction in women preeclampsia. The investigators hypothesise that in preeclampsia activated neutrophils may affect maternal immune system thus leading to myocardial injury and altered cardiac function. The study intends to identify the mechanisms by which the maternal immune system (focusing on neutrophil and T-cell subsets) affects cardiac function in women with preeclampsia. Specific aims to be addressed are:

Aim 1: To correlate specific neutrophil phenotype(s) and function to cardiac function in women with preeclampsia during pregnancy

Aim 2: To test whether specific activated neutrophil phenotype persists postpartum and whether this neutrophil phenotype correlates with cardiac function in women with preeclampsia postpartum

The study population will comprise of 3 groups:

1. Normotensive pregnant (~33 patients)
2. Pregnancy-induced hypertension (PIH; New-onset hypertension after 20 weeks without proteinuria; ~33 patients)
3. Preeclampsia (~34 patients)

Cardiac function will be evaluated using cardiovascular magnetic resonance, echocardiography and cardiac markers in the blood. The participants immune system will be assessed from blood samples looking at the immune cells, hormone levels and inflammatory and non-inflammatory mediators.

The secondary research objective is to investigate whether changes in the immune system and cardiac function in participants is persistent after delivery. Therefore participants will have scans and blood tests both antenatally and at 3 months postnatally.

By identifying key changes in immune cell type and function with cardiac abnormalities in women with preeclampsia, data obtained from this study could provide novel insight into how the maternal immune system influences cardiac changes in normal and preeclamptic pregnancies. Identifying such links could pave the way for future therapeutic targets.

DETAILED DESCRIPTION:
Study design

The overall aim of the clinical observational study is to determine whether the pro-inflammatory immune cell phenotype observed in women with preeclampsia (PE) can be correlated to cardiac function during and after pregnancy and in the postpartum period .

The study team will comprise of Dr Alice Christensen (PhD candidate), who will consent patients within the study group and carry out the clinical and laboratory aspects of the study; Dr Suchita Nadkarni (primary supervisor) who will oversee and train Dr Christensen on all basic science aspects of the study; Prof Steve Thornton and Dr Elena Greco (clinical supervisors) who will be the obstetric leads on the study; Consultant cardiologists will include Dr Neha Sekhri who will be primary contact for any cardiac issues, Dr Anna Herrey , who will oversee the analyses of imaging aspect of the study and Dr Kate Von Klemperer who will liaise with and advise Dr Christensen at both The Royal London and Barts Hospitals regarding echocardiography (echo). To this end, ~100 pregnant women will be recruited from The Royal London Hospital.

The study population will comprise of 3 groups:

1. Preeclamptic patients (34 patients)
2. Pregnancy-induced hypertension (PIH; 33 patients)
3. Healthy pregnant women (33)

Normotensive and PIH patients will be matched for gestational age with PE patients. Echocardiography and non-contrast cardiovascular magnetic resonance (CMR) studies will be carried out in all patients in the study upon enrolment and 3-months post partum, on the assumption that any physiological cardiovascular changes related to pregnancy will have resolved by then. Dr Anna Herrey - a leading expert in CMR in pregnant women will over-see the image analyses in the study. Dr Herrey has recently published a paper outlining the safety of carrying out CMR in pregnant women and the comparative resolution without the use of gadolinium contrast (Herrey et al 2019). Cardiac function will be assessed by echocardiography examination measuring ejection fraction, strain and diastolic function (as well as pulse wave velocity). Myocardial tissue characteristics will be assessed with non-contrast CMR (T1 and T2 mapping and full volumetric assessment, the gold standard for LV function analysis(Bellenger et al 2000 and Grothues et al 2002)). Any patient within the study group who demonstrates abnormal cardiac changes at 3-months post partum will be referred to Dr Sekhri for a 6-months follow-up (under NHS care at this time point). All cardiac scans will be carried out as an outpatient at Barts Hospital except for women with severe PE where the echocardiography will be carried out at bedside, upon admission to the ward. Thus, these women will not have CMR studies at enrolment but will be invited to attend the follow-up at 3 months for CMR and echocardiography studies.

Time- matched blood samples will be taken from patients to assess immune cell phenotypes. Plasma samples will be collected for the analyses of cardiac specific factors (BNP, troponin) as well as measurement of steroid hormones (progesterone and oestradiol), and soluble inflammatory and anti-inflammatory mediators. In order to limit bias within the study, all CMR image analyses (done by Dr Herrey) will be blinded. Dr Sekhri will be available for second reporting to assess interobserver variability of the CMR studies. Should any difference become apparent between early- and late-onset PE (PE which develops before and after 34 weeks gestation, respectively), sub-groups will be analysed within the PE group. This initial pilot study will inform power calculations for further studies in early and late onset disease.

Study procedures

Follow-up procedures

All patients recruited to the study, except those with severe PE, will be followed up as outpatients at The Royal London and will be asked to attend a hospital visit at Barts Hospital for CMR studies.

Participant withdrawal

Participants will have the option to submit a written request to be withdrawn from the trial at any stage. Participants will also have the option to withdraw consent from further participation in which circumstance no further data will be collected for inclusion. In the unfortunate event that a participant loses capacity, information gathered will continue to be used but no further data will be recorded.

The investigators will also ask participants if they can retain their contact information so that the investigators may contact them to take part in future research related to to current study. This request will be asked on the consent form.

End of Study Definition

The end of the study will be defined by achieving the proposed patient numbers per patient group (outlined above).

Statistical considerations

As this will be a pilot study the investigators cannot perform power calculations on the number of patients needed. the numbers for each patient group have been chosen based on the realistic numbers of patients that they believe can be recruited over the initial 1 year period and subsequent follow-up studies on these patients.

Method of analysis

With the support of our local NIHR bioinformatics and bio-repository facility (http://www.whri.qmul.ac.uk/core-facilities/nihr-bioinformatics-and-bio-repository), multiple parameters will be analysed using multiple group comparisons (ANOVAs) to increase power. In order to limit bias within the study, all CMR image analyses (done by Dr Herrey and Dr Sekhri) will be blinded, and interobserver variability will be measured.

The investigators will use flow cytometry to analyse immune cell phenotype. This is a well-established method. Dr Nadkarni's laboratory has access to a flow cytometry core facility, which has machines that can identify up 12 phenotypic markers on any given cell. Moreover, Dr Nadkarni, the Chief Investigator, and her group, have extensive experience in immune cell phenotyping using this method. The key advantages are:

1. It is the gold-standard for immune cell phenotyping
2. A minimal amount of blood are needed (max 200μls)
3. Antibodies are commercially available and have been extensively validated by ourselves and others
4. Dr Nadkarni has developed a high throughput method to analyse many samples at once, thereby minimising handling error

All samples will be processed an analysed within 1 hour of sample collection to minimise degradation of proteins on the surface of the immune cells.

The investigators also propose to look at circulating factors in the plasma and this will be carried out using commercially available ELISA kits.

The primary endpoint will be to determine whether there is a correlation between aberrant immune cell phenotypes and abnormal cardiac function within our preeclampsia patient cohort, compared to normal healthy and PIH groups. Furthermore, analyses will be carried out to find statistically significant cardiac functional and phenotypic differences between our preeclamptic and PIH patient cohorts, which will improve our understanding of cardiac function between the patient groups.

Ethics

Application for the current study is pending following submission. Informed consent will be obtained and recorded as described as above. Allowances for special groups are detailed above.

Incidental Findings

Should any incidental findings of clinical significance arise during the course of the study, the participants GP and clinical care team will be informed. Consent to contact the GP will be sought during the enrolment process.

Annual Safety Reporting

The CI will send an Annual Progress Report to the REC and the sponsor using the HRA template on the anniversary of the REC "favourable opinion".

Data management

All data generated will be stored within an Excel spreadsheet combining clinical and lab data. The spreadsheet will be password protected stored with a secure hard drive on a protected computer. Access to the password and data will be on a strict need-to-know basis. A full audit trail will be in place.

Source Data

Source data for this study will comprise of initial diagnoses of preeclampsia or pregnancy induced hypertension, which will be obtained from the obstetric care team, lead by Dr Elena Greco at the Royal London. These will be in the form of blood test results and/or scan images of the pregnancy.

Subsequent source data will be CMR images taken at the initial time point (diagnoses of preeclampsia and gestational age-matched controls) and follow-up CMR image data at the 2nd time point of the study (3 months post-partum). In addition to CMR images, source data will also be obtained from the laboratory phenotyping of blood samples taken from patients at the time points mentioned above.

Investigators who are directly involved with the study will have access to the source data. In some cases, where it is deemed best for the patient and their ongoing care, clinicians may seek advice from other experts, which may require their access to the source data.

Confidentiality

The investigators will undertake pseudorandomisation, whereby the patient is only be identifiable by their hospital number. As this will be a follow-up study, the investigators will need to link the patient and so this study will not be completely anonymised.

Record retention and archiving

The study data and documentation will be archived in accordance with the relevant regulatory requirements and site SOPs.

A unique alphanumeric patient identifier will be allocated to each participant at the start of the study. Data will be stored using the unique participant identifiers on a secure database. Data will not be stored on personal computers. Confidential documents will be stored in a locked cupboard located in a secure room. Clinical notes will be handled according to trust protocol. The Data Protection Act and the NHS confidentiality code of practice will be adhered to throughout this study. Data may be shared with members of the clinical team to allow ongoing clinical care.

GCP guidelines require that the investigator or the institution maintains all Case Report Forms and all source documents that support the data collected from each participant plus all trial documentation. Measures will be taken to prevent accidental or premature destruction of these documents. Essential documents must be retained for at least 20 years. It is the responsibility of the sponsor to inform the investigator when these documents no longer need to be retained. If the responsible investigator retires or leaves the institution responsibility for the documentation must be transferred to a person who will accept their custody

Sample preparation and collection

Blood samples to assess immune cell phenotypes will be collected from patients who have read the information sheet and signed the consent form. on the day of the cardiac MRI. A maximum volume of 15mls will be taken from the patient at any one time and collected into sodium citrate tubes.

Laboratory procedures

The majority of the blood samples will undergo phenotypic analyses using the flow cytometry method. Briefly, 50 microlitres of blood will be labelled with commercially-available antibodies that are conjugated to flurochromes that can be detected by lasers on the flow cytometer. Specialised software will enable the analyses of the assessment of phenotypic markers that are expressed on immune cells.

The samples will also be isolated for specific immune cell including neutrophils and T-cells, which will be stored in a secure -80oC freezer and may be subsequently used for genetic testing, including next generation and whole genome sequencing. Such deep sequencing will allow us to assess genetic changes that may occur alongside the phenotypic changes in the immune cells.

Plasma will also be collected from these samples to assess circulating factors, to be assessed by commercially-available kits.

Sample storage and transfer

Blood samples will be taken by the Research Fellow, Dr Alice Christensen, at Barts Heart Centre, where the Cardiac MRIs are to be carried out. Samples will be stored in an NHS fridge until transfer to laboratory. Barts Heart Centre is a maximum ten-minute walk to the William Harvey Research Institute where the laboratory is based. Samples will be transferred by Dr Christensen to the laboratory using secure sample transfer boxes to be brought to the laboratory. All blood samples will be processed within one hour of collection.

Safety reporting

Due to the observational nature and design of this study, safety reporting of adverse events will not occur.

Monitoring and auditing

The Sponsor or delegate retains the right to audit any study, study site or central facility. In addition, any part of the study may be audited by the funders where applicable.

On-site monitoring will be performed as per the study monitoring plan. Monitoring will include source data verification.

Monitoring of the centre may be undertaken by a trained study monitor or monitors, to verify the study documentation.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 years
* Singleton pregnancy
* Live fetus at 11-13 weeks of gestation
* Informed, written consent

Exclusion Criteria:

* Unwilling or unable to give consent
* Pre-eclamptic women with pre-existing conditions

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients attending The Royal London Hospital for antenatal care
Sampling Method: Non-Probability Sample
Enrollment: 86 (Actual)
Dates: Start 2020-01-07 (Actual); Primary Completion 2024-03-06 (Actual); Study Completion 2024-03-06 (Actual)

PRIMARY OUTCOMES:
Immune function and cardiac function in preeclampsia | 3 years
  To correlate maternal immune cell phenotype(s) and function to cardiac function in women with preeclampsia

SECONDARY OUTCOMES:
Postpartum immune function and cardiac function in preeclampsia | 3 years
  To investigate whether specific maternal immune cell phenotype(s) and altered cardiac function in women with PE persist in the post-partum period (up to 3 months after delivery).

CONTACTS AND LOCATIONS:
Overall Officials: Suchita Nadkarni, Study Director — Queen Mary University London
Locations (1):
- Barts Health NHS Trust, The Royal London Hospital, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Nadkarni S, Smith J, Sferruzzi-Perri AN, Ledwozyw A, Kishore M, Haas R, Mauro C, Williams DJ, Farsky SH, Marelli-Berg FM, Perretti M. Neutrophils induce proangiogenic T cells with a regulatory phenotype in pregnancy. Proc Natl Acad Sci U S A. 2016 Dec 27;113(52):E8415-E8424. doi: 10.1073/pnas.1611944114. Epub 2016 Dec 12. PMID 27956610
- [Background] Herrey AS, Francis JM, Hughes M, Ntusi NAB. Cardiovascular magnetic resonance can be undertaken in pregnancy and guide clinical decision-making in this patient population. Eur Heart J Cardiovasc Imaging. 2019 Mar 1;20(3):291-297. doi: 10.1093/ehjci/jey162. PMID 30462196
- [Background] Wenger NK. Recognizing pregnancy-associated cardiovascular risk factors. Am J Cardiol. 2014 Jan 15;113(2):406-9. doi: 10.1016/j.amjcard.2013.08.054. Epub 2013 Oct 6. PMID 24188889
- [Background] Bellenger NG, Davies LC, Francis JM, Coats AJ, Pennell DJ. Reduction in sample size for studies of remodeling in heart failure by the use of cardiovascular magnetic resonance. J Cardiovasc Magn Reson. 2000;2(4):271-8. doi: 10.3109/10976640009148691. PMID 11545126
- [Background] Grothues F, Smith GC, Moon JC, Bellenger NG, Collins P, Klein HU, Pennell DJ. Comparison of interstudy reproducibility of cardiovascular magnetic resonance with two-dimensional echocardiography in normal subjects and in patients with heart failure or left ventricular hypertrophy. Am J Cardiol. 2002 Jul 1;90(1):29-34. doi: 10.1016/s0002-9149(02)02381-0. PMID 12088775